CLINICAL TRIAL: NCT06959407
Title: Efficacy Of Oral Dexamethasone Versus Parenteral Dexamethasone In The Management Of Mild To Moderate Croup
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arooj Khan (Other)
Responsible Party: Sponsor-Investigator, Arooj Khan, Post Graduate Resident, Department of Child Health, Khyber Teaching Hospital
Organization: Khyber Teaching Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 410/DME/KMC
Record Dates: First submitted 2025-04-28; First posted 2025-05-06 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Laryngotracheobronchitis; Croup
MeSH Terms: conditions — Croup | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (oral dexamethasone ) (Active Comparator): Patients in group A will receive oral dexamethasone which will be administered at 0.6mg/kg as single dose
  Interventions: Drug: oral dexamethasone
- Group B (intramuscular dexamethasone ) (Active Comparator): Patients in group B will receive intramuscular dexamethasone which will be administered in 0.6mg/kg strength as intra-gluteal injection as single dose
  Interventions: Drug: intramuscular dexamethasone

INTERVENTIONS:
Drug: oral dexamethasone — Patients in group A will receive oral dexamethasone which will be administered at 0.6mg/kg as single dose
  Arms: Group A (oral dexamethasone )
Drug: intramuscular dexamethasone — Patients in group B will receive intramuscular dexamethasone which will be administered in 0.6mg/kg strength as intra-gluteal injection as single dose
  Arms: Group B (intramuscular dexamethasone )

SUMMARY:
Croup (laryngotracheobronchitis) is a viral infection of the upper airway that causes throat swelling, leading to a barking cough, stridor, and hoarseness. It mainly affects children aged 6 months to 12 years, peaking at around 2 years. Most cases are mild and self-limiting. Emergency treatments include cool mist, nebulized epinephrine, and steroids. Steroid therapy, particularly dexamethasone (oral or intramuscular), is commonly used, with recent studies suggesting intramuscular dexamethasone may be more effective. However, most research has focused on hospitalized patients, and there is a lack of local data for mild cases. This study aims to address that gap and improve patient counseling and future research

ELIGIBILITY:
Inclusion Criteria:

* Patient age 2 to 12 years
* Both genders
* Diagnosed with croup as operational definitions

Exclusion Criteria:

* Patients with chronic pulmonary disease like tuberculosis,
* Allergy or contraindication of corticosteroid (history of tuberous sclerosis, history of varicella infection during the past three weeks), to corticosteroids,
* history of corticosteroid administration during the last four weeks,
* foreign body
* patients with immunodeficiency disorder

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Settlement of symptoms of Croup | within 24 hours
  complete or partial settlement of symptoms i.e barking cough, inspiratory stridor, difficulty in breathing and hoarseness of voice.

CONTACTS AND LOCATIONS:
Locations (1):
- Khyber Teaching Hospital, Peshawar, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Smith DK, McDermott AJ, Sullivan JF. Croup: Diagnosis and Management. Am Fam Physician. 2018 May 1;97(9):575-580. PMID 29763253
- [Result] Parker CM, Cooper MN. Prednisolone Versus Dexamethasone for Croup: a Randomized Controlled Trial. Pediatrics. 2019 Sep;144(3):e20183772. doi: 10.1542/peds.2018-3772. Epub 2019 Aug 15. PMID 31416827
- [Result] Lin SC, Lin HW, Chiang BL. Association of croup with asthma in children: A cohort study. Medicine (Baltimore). 2017 Sep;96(35):e7667. doi: 10.1097/MD.0000000000007667. PMID 28858086
- [Result] Peltz A, Wu CL, White ML, Wilson KM, Lorch SA, Thurm C, Hall M, Berry JG. Characteristics of Rural Children Admitted to Pediatric Hospitals. Pediatrics. 2016 May;137(5):e20153156. doi: 10.1542/peds.2015-3156. Epub 2016 Apr 11. PMID 27244794
- [Result] Parikh K, Hall M, Mittal V, Montalbano A, Gold J, Mahant S, Wilson KM, Shah SS. Comparative Effectiveness of Dexamethasone versus Prednisone in Children Hospitalized with Asthma. J Pediatr. 2015 Sep;167(3):639-44.e1. doi: 10.1016/j.jpeds.2015.06.038. PMID 26319919